CLINICAL TRIAL: NCT04086680
Title: Use of the Idylla Platform for the Detection of EGFR Mutations in Liquid- Based Cytology Specimens of Lung Adenocarcinoma
Brief Title: The Detection of EGFR Mutations in Liquid Based Cytology Samples
Status: Completed | Type: Observational
Sponsor: Royal Cornwall Hospitals Trust (Other)
Collaborators: Biocartis NV (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019.RCHT.24
Record Dates: First submitted 2019-09-10; First posted 2019-09-11 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2019-06

CONDITIONS: Adenocarcinoma of Lung
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will investigate whether liquid based cytology specimens are a feasible alternative to formalin-fixed paraffin embedded histology samples for detection of epidermal growth factor receptor (EGFR) mutations in lung adenocarcinoma using the Biocartis Idylla platform. The Biocartis Idylla is a fully automated, real-time PCR based molecular diagnostics system. The Idylla carries out the entire analytical process from sample to result.

This study will be based in the cytology department at Royal Cornwall Hospital as part of a service improvement. It will use residual material from existing samples sent to the laboratory as part of the routine service. It will use existing material from patients diagnosed with lung adenocarcinoma by cytology using the current, validated procedure which uses formalin-fixed paraffin embedded (FFPE) samples over a 10 month period. EGFR mutation results obtained using the validated procedure (formalin fixed paraffin embedded) will be compared to those produced using liquid based cytology samples.

DETAILED DESCRIPTION:
The presence of activating epidermal growth factor receptor (EGFR) mutations identifies patients with lung adenocarcinoma in which EGFR tyrosine kinase inhibitors (TKI) can be a potential first-line treatment. The TKIs currently available are erlotinib, gefitinib and afatinib, which work by blocking receptor tyrosine kinase activity, thereby halting cell proliferation and causing cell death. Several studies have found that first-line TKI treatment prolongs progression free survival in comparison to standard chemotherapy, and is also associated with a more favourable tolerability and less adverse effects.

Samples for EGFR mutation analysis are collected from patients by endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) and bronchial brushings and washings. EBUS-TBNA provides a minimally invasive method for tissue sampling from radiologically suspicious lymph nodes in the chest using a fine-gauge needle. Samples obtained are collected and sent to the laboratory for processing. At present, laboratories rely on the use of formalin-fixed paraffin embedded (FFPE) samples for EGFR testing, therefore clots are produced in the laboratory using the collected tissue fragments. The clotted sample must then be fixed in formalin before being processed in the histology laboratory to produce slides for microscopic examination by the consultant pathologist. Once adenocarcinoma is diagnosed, FFPE samples are then sent for EGFR mutation analysis. The current laboratory process takes approximately 5 days.

Liquid based cytology (LBC) specimens obtained through the same sampling procedures are also prepared in the laboratory and fixed using a methanol based solution (PreservCyt). Previous research has been carried out to determine whether LBC samples can be used instead of FFPE samples for the detection of EGFR mutations with favourable results. Examples of this include research by Zhao et al (2017), Satouchi et al (2017), De Luca et al (2017) and Malapelle et al (2016). A switch to the use of LBC samples for EGFR testing would remove multiple processing steps in the sample pathway to mutation testing. Immunocytochemistry will be required in the majority of cases for confirmation of adenocarcinoma. This faster pathway would be beneficial in cases of already confirmed adenocarcinoma for second line EGFR treatment testing (T790M) and in cases where the residual cytology sample, that would normally be discarded, can be utilised for testing, optimising the potential of the sampling.

This study will investigate whether LBC specimens are a feasible alternative to FFPE samples for detection of EGFR mutations using the Biocartis Idylla platform.

If liquid based cytology samples are found to be a feasible alternative this could result in:

* Quicker turnaround time of results in cases of unequivocal adenocarcinoma. This would provide earlier access to TKIs allowing for optimal patient management.
* Easier sample preparation within the laboratory
* Would allow for efficient use of all material acquired from the sampling procedures. For example additional testing could be performed on the FFPE tissue in place of EGFR testing which could aid in diagnosis. Increase in efficient use of material could also prevent repeats of the EBUS procedure on patients.
* Methanol has been found to be a superior fixative than formalin. Use of liquid based cytology samples may allow for better results from molecular testing.
* Would provide support to the idea that molecular testing for other cancers may be able to be carried out on liquid based cytology samples for example BRAF mutation testing for melanoma. Also provides support of the use of other liquid samples for molecular testing such as blood samples which could be tested for circulating tumour cells (less invasive sampling).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lung adenocarcinoma by the cytology laboratory at Royal Cornwall Hospital Trust using the current, validated method on formalin-fixed paraffin embedded samples within the time period of the study. This will include both patients with wild type lung adenocarcinoma and also patients with lung adenocarcinoma with EGFR mutations.

Exclusion Criteria:

* Samples received by the cytology laboratory following the sampling procedures that are not diagnosed as lung adenocarcinoma during the time period of the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples from patients who have been diagnosed with lung adenocarcinoma by the cytology laboratory at Royal Cornwall Hospital Treliske using the current validated method on formalin-fixed paraffin embedded samples.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Significance of using liquid based cytology samples for EGFR mutation detection using the Idylla platform (in comparison to the use of FFPE samples) | 10 months
  The relative sensitivity and specificity will be calculated. Significance of use of liquid based cytology samples will be calculated using McNemars chi-squared test.

CONTACTS AND LOCATIONS:
Locations (1):
- Cytopathology Laboratory Royal Cornwall Hospital, Truro, Cornwall, United Kingdom